CLINICAL TRIAL: NCT01602562
Title: A Multicenter, Open-label Study to Evaluate Preventive Efficacy for Herpes Simplex Virus Infection and Safety of 256U87 (Valaciclovir Hydrochloride) in Adult and Pediatric Hematopoietic Stem Cell Transplantation Patients
Brief Title: Valaciclovir Hydrochloride Phase III for Hematopoietic Stem Cell Transplantation Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 116100
Record Dates: First submitted 2012-05-17; First posted 2012-05-21 (Estimated); Results first posted 2014-02-24 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-06

CONDITIONS: Herpes Simplex
Keywords: Herpes simplex infection; valaciclovir; herpes simplex virus; hematopoietic stem cell transplantation
MeSH Terms: conditions — Herpes Simplex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VACV (256U87; valaciclovir hydrochloride) (Experimental): Adult patients (16-65 years): A VACV tablet (containing 500mg of valaciclovir) is orally given twice daily. Pediatric patients (1-16 years): VACV granules are orally given at a dose of 25 mg/kg b.w. twice daily. The maximum dose per treatment is limited to 500 mg. Pediatric patients weighing 40 kg or over may be orally given a VACV tablet (containing 500 mg of valaciclovir) twice daily.
  Interventions: Drug: VACV tablets (Adults or pediatrics) or granules (pediatrics)

INTERVENTIONS:
Drug: VACV tablets (Adults or pediatrics) or granules (pediatrics) — A white to slightly yellowish white film coated tablet contains 556 mg of valaciclovir hydrochloride (500 mg of valaciclovir)). VACV granules have no or slightly specific odor.
  Other Names: 256U87 tablet or granule

SUMMARY:
The purpose of this study is to evaluate the preventive efficacy for HSV infection and safety of valaciclovir (VACV) in the adult and pediatric HSCT patients.

DETAILED DESCRIPTION:
This clinical study is a multicenter open-label study on the adult and pediatric hematopoietic stem cell transplantation (HSCT) patients. The primary objective is to confirm the preventive efficacy for herpes simplex virus (HSV) infection of 256U87 (VACV: valaciclovir) due to the treatment before or immediately after hematopoietic stem cell transplantation. The secondary objective is to confirm the safety of VACV in the case of its use for such a purpose.

This clinical study consists of the following two periods: the screening period lasting 7 days at the longest and the administration period from 7 days before HSCT to 35 days after HSCT (43 days in total). During the administration period, adult patients are orally given a VACV tablet twice daily, while pediatric patients are orally given VACV granules twice daily at a dose of 25 mg/kg b.w. (maximum dose per treatment: 500 mg). Pediatric patients weighing 40 kg or over may be orally given a VACV tablet twice daily.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are planning to undergo hematopoietic stem cell transplantation, except cord blood transplantation.
* Patients aged from 1 and above to under 65 at the time of informed consent.
* Patients who can submit their voluntary written informed consent if they are 12 years old and over.
* Patient is male or female. Male patients must be willing to use adequate contraception during the study. Female patients of childbearing potential must agree to consistently perform any of the contraceptive methods.
* QTc <450 msec, or QTc <480 msec in patients with bundle branch block. (values based on either single ECG values or triplicate ECG averaged QTc values)
* Liver test (aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <2x upper limit of normal (ULN); alkaline phosphatase (Al-P)and total bilirubin <=1.5xULN (total bilirubin >1.5xULN is acceptable if direct bilirubin <35%).

Exclusion Criteria:

* Patients with a history of HSCT.
* Patients who are judged to be in the following condition by the investigator (or subinvestigator): the clinical severity of malabsorption syndrome, vomiting, mucositis or other gastrointestinal dysfunction is so serious that orally administered VACV can not be absorbed.
* Patients who have known nucleoside analogs hypersensitivity.
* Patients who have a concurrent or past history of renal function disorder (serum creatinine >=1.5x ULN).
* Patients who have serious complication (eg, other malignant tumours, cardiac disorder, juvenile diabetes).
* Patients who are currently treated with the prohibited concomitant drugs.
* Patients with evidence of chronic hepatitis B or C.
* Patients with AIDS or patients infected with HIV.
* Patients who were given other trial products within 30 days before initiation of administration of this trial product or those who intend to participate in other clinical trials.
* Patients who are pregnant or probably pregnant.
* Patients who can not follow the protocol because of psychological, family, social or geological reasons.
* Patients are not allowed to participate in this clinical trial if the investigator (or subinvestigator) judges that their participation is inappropriate.

Ages: 1 Year to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2012-05-07; Primary Completion 2013-05-01 (Actual); Study Completion 2013-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- Japan (8):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 116100 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116100 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116100 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116100 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Adult Participants: VACV 500 mg Tablet: Adult participants (between 16 and 65 years of age) received a valaciclovir hydrochloride (VACV) tablet containing 500 milligrams (mg) of valaciclovir orally twice daily for 43 days, from 7 days before hematopoietic stem cell transplantation (HSCT) to 35 days after HSCT. A VACV tablet was administered once daily on Day -7 (7 days before HSCT) and on Day 35 (35 days after the final administration of HSCT).
- Pediatric Participants: VACV 500 mg Granules/Tablets: Pediatric participants (between 1 and <16 years of age) received VACV granules orally at a dose of 25 mg/kilogram (kg) body weight twice daily for 43 days, from 7 days before HSCT to 35 days after HSCT. The maximum dose per treatment was limited to 500 mg. Participants weighing 40 kg or more could have been given a VACV tablet (containing 500 mg of valaciclovir) orally twice daily. VACV granules were administered once daily on Day -7 (7 days before HSCT) and on Day 35 (35 days after the final administration of HSCT).
Period: Overall Study
Arm/Group | Adult Participants: VACV 500 mg Tablet | Pediatric Participants: VACV 500 mg Granules/Tablets
Started | 21 | 19
Completed | 16 | 16
Not Completed | 5 | 3
Not completed — Adverse Event | 3 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Adult Participants: VACV 500 mg Tablet: Adult participants (between 16 and 65 years of age) received a VACV tablet containing 500 mg of valaciclovir orally twice daily for 43 days, from 7 days before HSCT to 35 days after HSCT. A VACV tablet was administered once daily on Day -7 (7 days before HSCT) and on Day 35 (35 days after the final administration of HSCT).
- Pediatric Participants: VACV 500 mg Granules/Tablets: Pediatric participants (between 1 and <16 years of age) received VACV granules orally at a dose of 25 mg/kg body weight twice daily for 43 days, from 7 days before HSCT to 35 days after HSCT. The maximum dose per treatment was limited to 500 mg. Participants weighing 40 kg or more could have been given a VACV tablet (containing 500 mg of valaciclovir) orally twice daily. VACV granules were administered once daily on Day -7 (7 days before HSCT) and on Day 35 (35 days after the final administration of HSCT).
- Total: Total of all reporting groups
Arm/Group | Adult Participants: VACV 500 mg Tablet | Pediatric Participants: VACV 500 mg Granules/Tablets | Total
Number analyzed (Participants) | 21 | 19 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.6 (14.32) | 7.5 (4.69) | 29.1 (23.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 12 | 12 | 24
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - Japanese Heritage | 21 | 19 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Herpes Simplex Virus (HSV) Infection
Description: Viral isolation/identification was conducted if the investigator (or subinvestigator) suspected HSV infection according to the relevant clinical symptoms (oral mucositis, skin infection, genital herpes, and pneumonia). If the result of viral isolation/identification was positive, the participant concerned was defined as a case of HSV infection. For reference, a virus deoxyribonucleic acid (DNA) identification (PCR) was simultaneously performed.
Time Frame: From Day -7 (7 days before HSCT) to Day 35 (35 days after HSCT)
Population: Full Analysis Set (FAS): all participants who were given VACV more than once and who could provide data evaluable with respect to the occurrence of HSV infection.
Measure: Number; unit: Participants
Arm/Group | Adult Participants: VACV 500 mg Tablet | Pediatric Participants: VACV 500 mg Granules/Tablets
Number analyzed (Participants) | 21 | 19
Participants | 0 | 0
Statistical Analysis 1: Comparison: Adult Participants: VACV 500 mg Tablet; Test type: Superiority or Other; percentage of participants = 0.00, 95% CI 2-sided [0.00 to 16.11] — The estimated value reflects the percentage of participants with an HSV infection
Statistical Analysis 2: Comparison: Pediatric Participants: VACV 500 mg Granules/Tablets; Test type: Superiority or Other; percentage of participants = 0.00, 95% CI 2-sided [0.00 to 17.65] — The estimated value reflects the percentage of participants with an HSV infection

2. Secondary Outcome: Number of Participants With Any Adverse Event (AE) or Any Serious Adverse Event (SAE)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition, or is an event of possible drug-induced liver injury. Refer to the general AE/SAE module for a list of AEs and SAEs.
Time Frame: From Day -7 (7 days before HSCT) to Day 35 (35 days after HSCT)
Population: Safety Population: All participants who received VACV more than once.
Measure: Number; unit: Participants
Arm/Group | Adult Participants: VACV 500 mg Tablet | Pediatric Participants: VACV 500 mg Granules/Tablets
Number analyzed (Participants) | 21 | 19
Participants
  Any AE | 13 | 11
  Any SAE | 2 | 1

3. Secondary Outcome: Mean Alkaline Phosphatase (ALP), Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Creatine Phosphokinase (CPK), Gamma Glutamyl Transferase (GGT), and Lactate Dehydrogenase (LD) Values at Screening, Day 14, and Day 35
Description: Blood samples were collected for the measurement of ALP, ALT, AST, CPK, GGT, and LD at Screening, Day 14, and Day 35.
Time Frame: Screening (SCR), Day 14, and Day 35
Population: Safety Population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed for different parameters/at different time points, so the overall number of participants analyzed reflects everyone in the Safety Population.
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | Adult Participants: VACV 500 mg Tablet | Pediatric Participants: VACV 500 mg Granules/Tablets
Number analyzed (Participants) | 21 | 19
International units per liter (IU/L)
  ALP, SCR, n=21, 19 | 247.1 (105.09) | 598.8 (132.37)
  ALP, Day 14, n=18, 17 | 358.7 (206.04) | 456.7 (206.98)
  ALP, Day 35, n=16, 16 | 314.9 (111.65) | 519.9 (183.83)
  ALT, SCR, n=21, 19 | 23.7 (10.98) | 20.7 (12.55)
  ALT, Day 14, n=18, 17 | 53.2 (63.38) | 62.1 (84.64)
  ALT, Day 35, n=16, 16 | 58.9 (36.92) | 62.0 (76.59)
  AST, SCR, n=21, 19 | 23.2 (9.01) | 27.1 (9.62)
  AST, Day 14, n=18, 17 | 39.8 (39.82) | 35.0 (34.88)
  AST, Day 35, n=16, 16 | 45.1 (19.12) | 54.0 (48.96)
  CPK, SCR, n=21, 19 | 65.1 (70.37) | 72.0 (40.63)
  CPK, Day 14, n=18, 17 | 20.5 (9.88) | 27.4 (28.85)
  CPK, Day 35, n=16, 16 | 42.1 (26.74) | 38.4 (26.48)
  GGT, SCR, n=21, 19 | 47.2 (34.94) | 24.8 (24.74)
  GGT, Day 14, n=18, 17 | 118.4 (113.63) | 27.5 (10.61)
  GGT, Day 35, n=16, 16 | 90.3 (70.96) | 50.7 (43.34)
  LD, SCR, n=21, 19 | 251.8 (179.06) | 213.3 (77.51)
  LD, Day 14, n=18, 17 | 215.4 (68.15) | 210.6 (103.09)
  LD, Day 35, n=16, 16 | 256.7 (65.92) | 255.9 (92.84)

4. Secondary Outcome: Mean Direct Bilirubin, Total Bilirubin, Creatinine, and Uric Acid Values at Screening, Day 14, and Day 35
Description: Blood samples were collected for the measurement of direct bilirubin, total bilirubin, creatinine, and uric acid at Screening, Day 14, and Day 35.
Time Frame: Screening (SCR), Day 14, and Day 35
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Micromoles per liter (µmol/L)
Arm/Group | Adult Participants: VACV 500 mg Tablet | Pediatric Participants: VACV 500 mg Granules/Tablets
Number analyzed (Participants) | 21 | 19
Micromoles per liter (µmol/L)
  Direct bilirubin, SCR, n=21, 19 | 2.931 (1.8843) | 2.970 (1.8769)
  Direct bilirubin, Day 14, n=18, 17 | 7.410 (11.5234) | 3.923 (3.0688)
  Direct bilirubin, Day 35, n=16, 16 | 2.351 (0.8550) | 2.565 (1.2488)
  Total bilirubin, SCR, n=21, 19 | 8.224 (5.4242) | 8.190 (3.9728)
  Total bilirubin, Day 14, n=18, 17 | 12.540 (14.8264) | 9.858 (8.6251)
  Total bilirubin, Day 35, n=16, 16 | 6.306 (1.9466) | 6.733 (3.1512)
  Creatinine, SCR, n=21, 19 | 62.6798 (19.71123) | 30.1025 (10.12416)
  Creatinine, Day 14, n=18, 17 | 46.7047 (16.31214) | 25.5320 (12.84039)
  Creatinine, Day 35, n=16, 16 | 58.7860 (18.83010) | 33.3710 (19.49749)
  Uric acid, SCR, n=21, 19 | 276.1571 (80.38764) | 259.5206 (63.88405)
  Uric acid, Day 14, n=18, 17 | 133.1691 (62.35442) | 137.5038 (56.34464)
  Uric acid, Day 35, n=16, 16 | 255.0205 (96.37167) | 238.6635 (101.47400)

5. Secondary Outcome: Mean Cholesterol, Chloride, Glucose, Potassium, Sodium, Triglyceride, and Urea/Blood Urea Nitrogen (BUN) Values at Screening, Day 14, and Day 35
Description: Blood samples were collected for the measurement of cholesterol, chloride, glucose, potassium, sodium, triglycerides, and urea/BUN at Screening, Day 14, and Day 35.
Time Frame: Screening (SCR), Day 14, and Day 35
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Groups:
- Pediatric Participants: VACV 500 mg Granules/Tablets: Pediatric participants (between 1 and & <16 years of age) received VACV granules orally at a dose of 25 mg/kg body weight twice daily for 43 days, from 7 days before HSCT to 35 days after HSCT. The maximum dose per treatment was limited to 500 mg. Participants weighing 40 kg or more could have been given a VACV tablet (containing 500 mg of valaciclovir) orally twice daily. VACV granules were administered once daily on Day -7 (7 days before HSCT) and on Day 35 (35 days after the final administration of HSCT).
Arm/Group | Adult Participants: VACV 500 mg Tablet | Pediatric Participants: VACV 500 mg Granules/Tablets
Number analyzed (Participants) | 21 | 19
Millimoles per liter (mmol/L)
  Cholesterol, SCR, n=21, 19 | 4.8149 (1.33518) | 4.1703 (0.70625)
  Cholesterol, Day 14, n=18, 17 | 4.0255 (1.06483) | 3.5504 (1.25610)
  Cholesterol, Day 35, n=16, 16 | 5.5324 (1.45536) | 4.1279 (1.01828)
  Chloride, SCR, n=21, 19 | 105.2 (2.83) | 103.3 (2.21)
  Chloride, Day 14, n=18, 17 | 104.4 (4.06) | 105.0 (2.06)
  Chloride, Day 35, n=16, 16 | 106.0 (2.99) | 104.0 (2.31)
  Glucose, SCR, n=21, 19 | 5.8127 (1.38621) | 6.0214 (1.83355)
  Glucose, Day 14, n=18, 17 | 7.2656 (2.31056) | 6.0996 (2.13721)
  Glucose, Day 35, n=16, 16 | 6.4808 (1.35160) | 5.7800 (1.41869)
  Potassium, SCR, n=21, 19 | 4.08 (0.402) | 4.01 (0.283)
  Potassium, Day 14, n=18, 17 | 3.93 (0.457) | 4.34 (0.449)
  Potassium, Day 35, n=16, 16 | 4.31 (0.521) | 4.09 (0.359)
  Sodium, SCR, n=21, 19 | 142.0 (1.92) | 140.2 (1.92)
  Sodium, Day 14, n=18, 17 | 140.3 (4.16) | 139.2 (1.55)
  Sodium, Day 35, n=16, 16 | 141.8 (2.29) | 139.3 (1.39)
  Triglycerides, SCR, n=21, 19 | 2.0760 (1.30955) | 1.3489 (0.75044)
  Triglycerides, Day 14, n=18, 17 | 1.8789 (0.95581) | 1.4185 (1.02762)
  Triglycerides, Day 35, n=16, 16 | 2.9486 (1.49324) | 1.6646 (1.04585)
  Urea/BUN, SCR, n=21, 19 | 4.2721 (1.61486) | 3.6903 (0.93331)
  Urea/BUN, Day 14, n=18, 17 | 4.8274 (3.76473) | 3.1332 (1.35997)
  Urea/BUN, Day 35, n=16, 16 | 3.7619 (1.72437) | 4.1657 (1.99412)

6. Secondary Outcome: Mean Albumin and Total Protein Values at Screening, Day 14, and Day 35
Description: Blood samples were collected for the measurement of albumin and total protein at Screening, Day 14, and Day 35.
Time Frame: Screening (SCR), Day 14, and Day 35
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Grams per liter (G/L)
Arm/Group | Adult Participants: VACV 500 mg Tablet | Pediatric Participants: VACV 500 mg Granules/Tablets
Number analyzed (Participants) | 21 | 19
Grams per liter (G/L)
  Albumin, SCR, n=21, 19 | 41.0 (3.07) | 41.5 (2.04)
  Albumin, Day 14, n=18, 17 | 34.6 (3.87) | 39.1 (3.04)
  Albumin, Day 35, n=16, 16 | 40.8 (3.34) | 40.9 (3.02)
  Total protein, SCR, n=21, 19 | 64.2 (5.83) | 66.2 (5.34)
  Total protein, Day 14, n=18, 17 | 57.6 (5.76) | 62.7 (5.08)
  Total protein, Day 35, n=16, 16 | 62.9 (4.75) | 65.3 (5.84)

7. Secondary Outcome: Mean Basophil, Eosinophil, Lymphocyte, Monocyte, and Total Neutrophil Values at Screening, Day 14, and Day 35
Description: Blood samples were collected for the measurement of basophils, eosinophils, lymphocytes, monocytes, and total neutrophils at Screening, Day 14, and Day 35.
Time Frame: Screening (SCR), Day 14, and Day 35
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of cells in blood
Arm/Group | Adult Participants: VACV 500 mg Tablet | Pediatric Participants: VACV 500 mg Granules/Tablets
Number analyzed (Participants) | 21 | 19
Percentage of cells in blood
  Basophils, SCR, n=21,19 | 1.05 (1.473) | 0.49 (0.470)
  Basophils, Day 14, n=16, 16 | 0.69 (1.661) | 0.14 (0.352)
  Basophils, Day 35, n=16, 15 | 1.09 (0.903) | 0.59 (0.380)
  Eosinophils, SCR, n=21, 19 | 3.67 (4.754) | 2.06 (1.974)
  Eosinophils, Day 14, n=16, 16 | 0.79 (2.770) | 0.59 (1.517)
  Eosinophils, Day 35, n=16, 15 | 4.10 (2.672) | 7.51 (10.357)
  Lymphocytes, SCR, n=21,19 | 32.72 (16.104) | 38.94 (21.616)
  Lymphocytes, Day 14, n=16, 16 | 13.61 (8.897) | 16.73 (17.909)
  Lymphocytes, Day 35, n=16, 15 | 37.08 (15.496) | 30.85 (20.338)
  Monocytes, SCR, n=21,19 | 7.90 (3.337) | 10.99 (7.565)
  Monocytes, Day 14, n=16, 16 | 15.32 (7.263) | 17.33 (12.061)
  Monocytes, Day 35, n=16, 15 | 14.54 (6.609) | 13.33 (7.021)
  Total neutrophils, SCR, n=21,19 | 54.46 (15.003) | 47.52 (22.667)
  Total neutrophils, Day 14, n=16, 16 | 63.53 (18.117) | 62.21 (23.273)
  Total neutrophils, Day 35, n=16, 15 | 42.76 (13.336) | 47.63 (20.745)

8. Secondary Outcome: Mean Platelet Count and White Blood Cell (WBC) Count at Screening, Day 14, and Day 35
Description: Blood samples were collected for the measurement of platelet count and WBC count at Screening, Day 14, and Day 35.
Time Frame: Screening (SCR), Day 14, and Day 35
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: giga (10^9) per liter (GI/L)
Arm/Group | Adult Participants: VACV 500 mg Tablet | Pediatric Participants: VACV 500 mg Granules/Tablets
Number analyzed (Participants) | 21 | 19
giga (10^9) per liter (GI/L)
  Platelet count, SCR, n=21,19 | 190.2 (126.32) | 167.7 (98.15)
  Platelet count, Day 14, n=18, 17 | 40.3 (20.73) | 58.2 (37.41)
  Platelet count, Day 35, n=16, 16 | 139.4 (79.29) | 119.0 (89.31)
  WBC count, SCR, n=21,19 | 4.01 (1.842) | 3.03 (1.873)
  WBC count, Day 14, n=16, 12 | 3.46 (2.955) | 2.23 (2.403)
  WBC count, Day 35, n=16, 14 | 5.00 (3.524) | 3.71 (2.189)

9. Secondary Outcome: Mean Red Blood Cell Count at Screening, Day 14, and Day 35
Description: Blood samples were collected for the measurement of the red blood cell count at Screening, Day 14, and Day 35.
Time Frame: Screening (SCR), Day 14, and Day 35
Population: Safety Population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the Safety Population.
Measure: Mean (Standard Deviation); unit: tera (10^12) per liter (TI/L)
Arm/Group | Adult Participants: VACV 500 mg Tablet | Pediatric Participants: VACV 500 mg Granules/Tablets
Number analyzed (Participants) | 21 | 19
tera (10^12) per liter (TI/L)
  SCR, n=21,19 | 3.165 (0.7583) | 3.293 (0.6529)
  Day 14, n=18, 17 | 2.932 (0.3479) | 2.908 (0.3854)
  Day 35, n=16, 16 | 3.297 (0.5021) | 3.073 (0.4797)

10. Secondary Outcome: Mean Hemoglobin Values at Screening, Day 14, and Day 35
Description: Blood samples were collected for the measurement of hemoglobin at Screening, Day 14, and Day 35.
Time Frame: Screening (SCR), Day 14, and Day 35
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Grams per liter (G/L)
Arm/Group | Adult Participants: VACV 500 mg Tablet | Pediatric Participants: VACV 500 mg Granules/Tablets
Number analyzed (Participants) | 21 | 19
Grams per liter (G/L)
  SCR, n=21,19 | 101.6 (24.84) | 99.3 (17.94)
  Day 14, n=18, 17 | 91.6 (10.02) | 85.1 (12.10)
  Day 35, n=16, 16 | 106.5 (16.36) | 94.4 (15.23)

11. Secondary Outcome: Number of Participants With the Indicated Result for the Indicated Urinalysis Parameters Tested by Dipstick at Screening, Day 14, and Day 35
Description: Urinalysis parameters included: urine bilirubin (UB), urine occult blood (UOB), urine glucose (UG), urine ketones (UK), urine protein (UP), and urine urobilinogen (UUG). The dipstick is a strip used to detect the presence or absence of these parameters in the urine sample. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameters can be read as negative (Neg), Trace, 1+, 2+, and 3+ (in order of increasing levels). Data are reported as the number of participants who had Neg, Trace, 1+, 2+, and 3+ levels at Screening, Day 14, and Day 35. If a category has not been reported for a specific parameter, then no participants were measured in that category.
Time Frame: Screening (SCR), Day 14, and 35
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Adult Participants: VACV 500 mg Tablet | Pediatric Participants: VACV 500 mg Granules/Tablets
Number analyzed (Participants) | 21 | 19
Participants
  UB, Neg, SCR, n=21, 19 | 21 | 19
  UB, Neg, Day 14, n=18, 17 | 18 | 17
  UB, Neg, Day 35, n=16, 16 | 16 | 16
  UOB, Neg, SCR, n=21, 19 | 19 | 19
  UOB, 2+, SCR, n=21, 19 | 2 | 0
  UOB, Neg, Day 14, n=18, 17 | 14 | 14
  UOB, Trace, Day 14, n=18, 17 | 2 | 2
  UOB, 1+, Day 14, n=18, 17 | 2 | 0
  UOB, 3+, Day 14, n=18, 17 | 0 | 1
  UOB, Neg, Day 35, n=16, 16 | 12 | 16
  UOB, Trace, Day 35, n=16, 16 | 1 | 0
  UOB, 1+, Day 35, n=16, 16 | 2 | 0
  UOB, 3+, Day 35, n=16, 16 | 1 | 0
  UG, Neg, SCR, n=21, 19 | 19 | 19
  UG, Trace, SCR, n=21, 19 | 2 | 0
  UG, Neg, Day 14, n=18, 17 | 14 | 17
  UG, Trace, Day 14, n=18, 17 | 1 | 0
  UG, 1+, Day 14, n=18, 17 | 1 | 0
  UG, 2+, Day 14, n=18, 17 | 1 | 0
  UG, 3+, Day 14, n=18, 17 | 1 | 0
  UG, Neg, Day 35, n=16, 16 | 15 | 16
  UG, Trace, Day 35, n=16, 16 | 1 | 0
  UK, Neg, SCR, n=21, 19 | 21 | 19
  UK, Neg, Day 14, n=18, 17 | 17 | 17
  UK, 1+, Day 14, n=18, 17 | 1 | 0
  UK, Neg, Day 35, n=16, 16 | 16 | 15
  UK, 1+, Day 35, n=16, 16 | 0 | 1
  UP, Neg, SCR, n=21, 19 | 19 | 14
  UP, Trace, SCR, n=21, 19 | 0 | 4
  UP, 1+, SCR, n=21, 19 | 0 | 1
  UP, 2+, SCR, n=21, 19 | 2 | 0
  UP, Neg, Day 14, n=18, 17 | 9 | 12
  UP, Trace, Day 14, n=18, 17 | 5 | 4
  UP, 1+, Day 14, n=18, 17 | 2 | 0
  UP, 2+, Day 14, n=18, 17 | 2 | 1
  UP, Neg, Day 35, n=16, 16 | 13 | 13
  UP, Trace, Day 35, n=16, 16 | 2 | 1
  UP, 1+, Day 35, n=16, 16 | 1 | 2
  UUG, Trace, SCR, n=21, 19 | 19 | 19
  UUG, 2+, SCR, n=21, 19 | 2 | 0
  UUG, Trace, Day 14, n=18, 17 | 17 | 15
  UUG, 1+, Day 14, n=18, 17 | 1 | 0
  UUG, 2+, Day 14, n=18, 17 | 0 | 1
  UUG, 3+, Day 14, n=18, 17 | 0 | 1
  UUG, Trace, Day 35, n=16, 16 | 16 | 15
  UUG, 3+, Day 35, n=16, 16 | 0 | 1

12. Secondary Outcome: Mean Urine Specific Gravity Values at Screening, Day 14, and Day 35
Description: Safety Population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the Safety Population.
Time Frame: Screening (SCR), Day 14, and Day 35
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Adult Participants: VACV 500 mg Tablet | Pediatric Participants: VACV 500 mg Granules/Tablets
Number analyzed (Participants) | 21 | 19
ratio
  SCR, n=21, 19 | 1.0146 (0.00705) | 1.0188 (0.00912)
  Day 14, n=18, 17 | 1.0158 (0.00628) | 1.0155 (0.00685)
  Day 35, n=16, 16 | 1.0137 (0.00572) | 1.0153 (0.00642)

13. Secondary Outcome: Change From Baseline in Systolic Blood Pressure and Diastolic Blood Pressure at Days 0, 7, 14, 21, and 35
Description: Blood pressure measurement included systolic blood pressure (SBP) and diastolic blood pressure (DBP). Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Days 0, 7, 14, 21, and 35
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Adult Participants: VACV 500 mg Tablet | Pediatric Participants: VACV 500 mg Granules/Tablets
Number analyzed (Participants) | 21 | 19
Millimeters of mercury
  SBP, Day 0, n=21, 19 | -1.8 (18.23) | -4.7 (16.85)
  SBP, Day 7, n=19, 17 | 0.9 (18.88) | -6.1 (16.34)
  SBP, Day 14, n=18, 17 | 4.3 (20.68) | -7.6 (18.61)
  SBP, Day 21, n=17, 17 | -1.4 (14.98) | -7.0 (13.88)
  SBP, Day 35, n=16, 16 | 2.8 (20.14) | -4.5 (15.08)
  DBP, Day 0, n=21, 19 | -2.7 (16.04) | -1.8 (13.63)
  DBP, Day 7, n=19, 17 | 1.6 (16.37) | 0.3 (13.87)
  DBP, Day 14, n=18, 17 | 3.4 (18.29) | -5.9 (14.69)
  DBP, Day 21, n=17, 17 | 1.5 (11.41) | -1.2 (11.91)
  DBP, Day 35, n=16, 16 | 4.7 (14.74) | -1.1 (11.20)

14. Secondary Outcome: Change From Baseline in Heart Rate at Days 0, 7, 14, 21, and 35
Description: Heart rate is defined as the number of heartbeats per unit of time. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Days 0, 7, 14, 21, and 35
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Adult Participants: VACV 500 mg Tablet | Pediatric Participants: VACV 500 mg Granules/Tablets
Number analyzed (Participants) | 21 | 19
Beats per minute
  Day 0, n=21, 19 | 1.1 (13.66) | -1.0 (17.15)
  Day 7, n=19, 17 | 13.3 (14.41) | 3.8 (20.42)
  Day 14, n=18, 17 | 12.5 (14.70) | 3.6 (25.47)
  Day 21, n=17, 17 | 16.4 (14.54) | 1.8 (21.14)
  Day 35, n=16, 16 | 19.2 (18.99) | 3.6 (23.60)

15. Secondary Outcome: Number of Participants With the Indicated Electrocardiogram (ECG) Findings at Screening and Day 35
Description: The number of participants with normal, abnormal - clinically significant (CS), and abnormal - not clinically significant (NCS) ECG findings, as well as the number of participants with no results (NR), at Screening and Day 35 are presented. Findings were determined to be normal, abnormal CS, and NCS by the investigator.
Time Frame: Screening (SCR) and Day 35
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | Adult Participants: VACV 500 mg Tablet | Pediatric Participants: VACV 500 mg Granules/Tablets
Number analyzed (Participants) | 21 | 19
Participants
  SCR, Normal, n=21, 19 | 16 | 19
  SCR, NCS, n=21, 19 | 5 | 0
  SCR, CS, n=21, 19 | 0 | 0
  SCR, NR, n=21, 19 | 0 | 0
  Day 35, Normal, n=16, 16 | 15 | 13
  Day 35, NCS, n=16, 16 | 1 | 2
  Day 35, CS, n=16, 16 | 0 | 0
  Day 35, NR, n=16, 16 | 0 | 1

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study medication until the end of the treatment (up to Day 43).
Description: SAEs and non-serious AEs are reported for members of the Safety Population, comprised of all participants who received VACV more than once.
Arm/Group | Adult Participants: VACV 500 mg Tablet | Pediatric Participants: VACV 500 mg Granules/Tablets
Serious Adverse Events (participants affected / at risk) | 2/21 | 1/19
Other Adverse Events (participants affected / at risk) | 13/21 | 11/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adult Participants: VACV 500 mg Tablet (N=21) | Pediatric Participants: VACV 500 mg Granules/Tablets (N=19)
Liver injury (Hepatobiliary disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adult Participants: VACV 500 mg Tablet (N=21) | Pediatric Participants: VACV 500 mg Granules/Tablets (N=19)
Diarrhoea (Gastrointestinal disorders) | 8 | 4
Nausea (Gastrointestinal disorders) | 5 | 3
Vomiting (Gastrointestinal disorders) | 3 | 5
Stomatitis (Gastrointestinal disorders) | 4 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 3
Constipation (Gastrointestinal disorders) | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Proctalgia (Gastrointestinal disorders) | 2 | 0
Tongue coated (Gastrointestinal disorders) | 0 | 2
Anal fissure (Gastrointestinal disorders) | 1 | 0
Anorectal discomfort (Gastrointestinal disorders) | 1 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Gastrointestinal mucosal disorder (Gastrointestinal disorders) | 0 | 1
Gingival swelling (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0
Oral discomfort (Gastrointestinal disorders) | 1 | 0
Oral disorder (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1
Parotid gland enlargement (Gastrointestinal disorders) | 1 | 0
Periproctitis (Gastrointestinal disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 7 | 2
Fluid retention (Metabolism and nutrition disorders) | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 3
Leukopenia (Blood and lymphatic system disorders) | 0 | 4
Neutropenia (Blood and lymphatic system disorders) | 0 | 3
Lymphopenia (Blood and lymphatic system disorders) | 0 | 2
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Xeroderma (Skin and subcutaneous tissue disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2
Bacteraemia (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 1 | 1
Acute sinusitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0
Molluscum contagiosum (Infections and infestations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 4
Aspartate aminotransferase increased (Investigations) | 1 | 4
Amylase increased (Investigations) | 0 | 3
Blood bilirubin increased (Investigations) | 2 | 1
C-reactive protein increased (Investigations) | 0 | 3
Blood urine present (Investigations) | 0 | 2
Hepatic enzyme increased (Investigations) | 2 | 0
Occult blood (Investigations) | 0 | 2
Antithrombin III decreased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Blood magnesium decreased (Investigations) | 1 | 0
Blood potassium decreased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 0 | 1
Blood sodium increased (Investigations) | 1 | 0
Glucose urine present (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 1 | 0
Red blood cell count decreased (Investigations) | 1 | 0
Urine output decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 1 | 0
Fatigue (General disorders) | 5 | 2
Pyrexia (Investigations) | 2 | 3
Chest pain (General disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Feeling abnormal (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 2
Dysgeusia (Nervous system disorders) | 1 | 0
Head discomfort (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Sensory disturbance (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 4 | 0
Delirium (Psychiatric disorders) | 1 | 0
Diplopia (Eye disorders) | 1 | 0
Dry eye (Eye disorders) | 0 | 1
Eye pruritus (Eye disorders) | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 1
Hypertonic bladder (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Liver injury (Hepatobiliary disorders) | 1 | 0
Bone marrow transplant rejection (Immune system disorders) | 1 | 0
Graft versus host disease in skin (Immune system disorders) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.